CLINICAL TRIAL: NCT01500954
Title: Microarray Analysis of microRNA Expression Profiles in Cutaneous Squamous Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Michael Sand, Principal Investigator, Ruhr University of Bochum
Other Study IDs: microRNA7
Record Dates: First submitted 2011-12-23; First posted 2011-12-29 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Cutaneous Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cutaneous squamous cell carcinoma (SCC) non.lesional skin
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- squamous cell carcinoma
- non-lesional skin

SUMMARY:
MicroRNAs (miRNAs) are a novel class of short RNAs which have shown to be dysregulated in a variety of cancers. Data of miRNA expression in cutaneous squamous cell carcinoma (cSCC) is very limited and microarray based genome wide miRNA expression profiles of cSCC have not been investigated so far.

DETAILED DESCRIPTION:
Patients with cutaneous SCC were enrolled in the present study. Tumor biopsies were taken from the center of the tumor. Adjacent healthy skin was biopsied as a control (intraindividual control). miRNA expression profiles of specimen were detected by microarray miRNA expression profiling. Microarray results were confirmed by TaqMan real-time quantitative polymerase chain reaction (RT-PCR).

ELIGIBILITY:
Inclusion Criteria:

* cutaneous squamous cell carcinoma

Exclusion Criteria:

* other skin cancer than cutaneous squamous cell carcinoma

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cutaneous squamous cell carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Falk G Bechara, PD Dr., Study Director — Department of Dermatology, Venereology and Allergology, Dermatologic Surgery Unit, Ruhr-University Bochum; Peter Altmeyer, Prof. Dr., Study Chair — Department of Dermatology, Venereology and Allergology, Ruhr-University Bochum; Michael Sand, Dr., Principal Investigator — Department of Dermatology, Venereology and Allergology, Dermatologic Surgery Unit, Ruhr-University Bochum
Locations (1):
- Department of Dermatology, Venereology and Allergology, Dermatologic Surgery Unit, Ruhr-University Bochum, Bochum, North Rhine-Westphalia, Germany

REFERENCES:
- [Result] Sand M, Skrygan M, Georgas D, Sand D, Hahn SA, Gambichler T, Altmeyer P, Bechara FG. Microarray analysis of microRNA expression in cutaneous squamous cell carcinoma. J Dermatol Sci. 2012 Dec;68(3):119-26. doi: 10.1016/j.jdermsci.2012.09.004. Epub 2012 Sep 13. PMID 23026055